CLINICAL TRIAL: NCT04200287
Title: Pilot Study to Improve Survivorship Care Related to Fertility and Family-building After Cancer
Brief Title: Study to Improve Survivorship Care Related to Fertility and Family-building After Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-52372; VAR0192 (Other: OnCore)
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Young adult female (YA-F) cancer survivors (Experimental): YA-F cancer survivors will complete a baseline survey (T1) of sociodemographic and patient reported outcomes (PRO) and then will be sent a link to access the decision aid tool (website) with instructions to review the website before their upcoming visit. A follow-up survey (T2) will be emailed 4-weeks post-baseline, prior to their clinic visit, to evaluate website access and PROs. A post-visit survey (T3) will be emailed 6- weeks post-baseline (after their survivorship care visit) to assess PROs.
  Interventions: Behavioral: Online decision aid tool

INTERVENTIONS:
Behavioral: Online decision aid tool — The decision aid intervention will be presented via a website

SUMMARY:
The goal of this research is to explore how a patient decision aid tool (website) given to patients prior to their survivorship care visits, may impact patient-provider communication about fertility and family-building after cancer; and assess the impact of using the tool on patient reported outcomes. The overall purpose of this research is to improve survivorship care by establishing a multi-disciplinary approach to managing cancer and fertility issues and prompt early referral to supportive and medical care resources.

DETAILED DESCRIPTION:
Objective 1: Establish feasibility and acceptability of conducting research with YA-F cancer survivors at the Stanford Cancer Institute (SCI) and Lucile Packard Children's Hospital (LPCH).

Hypothesis 1: Study procedures will be feasible in the given timeframe and acceptable to patients, as evidence by recruitment, enrollment, and completion rates and participant feedback.

Objective 2: Evaluate the impact of using the tool as a part of survivorship care on patient reported outcomes (PROs; i.e., information needs, fertility distress, decision-making uncertainty, and satisfaction with care).

Hypothesis 2: In a single-arm pilot study (N=20), use of the decision aid tool will lead to improvements in fertility distress, decision-making uncertainty, and satisfaction with care.

ELIGIBILITY:
Inclusion Criteria:

* completed cancer treatment at least 6-months prior, excluding long-term adjuvant or maintenance therapies
* report an interest in discussing fertility/family-building with a provider
* understands verbal and written English
* access to the Internet and use of a computer, tablet, or smartphone
* has a scheduled cancer survivorship visit within the study time frame

Exclusion Criteria:

* Prior hospitalization for a mental disorder or history of psychosis

Note: Survivors on adjuvant maintenance or endocrine treatment, such as tamoxifen, will not be excluded because clinical guidelines allow treatment delay or hiatus to accommodate fertility

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-09-11 (Actual); Study Completion 2021-09-11 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict Scale (DCS) | 6 weeks
  The Decisional Conflict Scale (DCS) is a validated survey that assesses personal uncertainty in making healthcare decisions; modifiable factors contributing to uncertainty; and the quality of the decision made. It is reliable and responsive to change, and the most widely used measure of decision-making quality. The survey has 16 questions, with responses on a 5-point scale ranging from "strongly agree" (1) to "strongly disagree" (5).
  Total scores range from 16 to 80, with higher scores indicating greater uncertainty (worse outcome). The outcome will be reported as the mean difference from baseline to 4-week and 6-week follow-up time points, with standard deviation.

SECONDARY OUTCOMES:
Unmet Fertility Information | 6 weeks
  This investigator-designed survey assesses perceived information needs about fertility topics such as the risk of infertility; risk of early menopause; options to assess fertility status; options to preserve fertility; and options for alternative family-building. The survey has 5 questions, each answered by a Yes / No response. Yes is scored as 1, and no is scored as 0. Total scores range from 0 to 5, with higher scores indicating greater perceived knowledge. The outcome will be reported as the mean difference from baseline to 4-week and 6-week follow-up time points, with standard deviation.
Reproductive Concerns After Cancer (RCAC) Scale | 6 weeks
  The Reproductive Concerns After Cancer (RCAC) Scale is a validated survey of cancer survivors' fertility and health concerns. The survey has 18 questions, answered on a 5-point scale ranging from "strongly disagree" (1) to "strongly agree" (5). Total scores range from 18 to 90, with higher scores indicating greater distress (worse outcome). The outcome will be reported as the mean difference from baseline to 4-week and 6-week followup time points, with standard deviation.
COMRADE | 6 weeks
  The COMRADE is a measure of patient-based outcomes of risk communication within patient-provider interactions and treatment decision-making effectiveness. It consists of two subscales: Satisfaction with Communication & Confidence in Decision-making. Items were adapted to refer to fertility and reproductive health care options. The measure has 20 questions. Items are answered on a 5-point scale from "Strongly Disagree" to "Strongly Agree," with high scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Benedict, Principal Investigator — Stanford University
Locations (1):
- Stanford Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT04200287/ICF_001.pdf